CLINICAL TRIAL: NCT04388085
Title: Validity, Reliability and Responsiveness of King's Sarcoidosis Questionnaire in a Danish Population
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SAR2
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-05

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The King's Sarcoidosis Questionnaire (KSQ) is a brief questionnaire assessing health status in patients with sarcoidosis. The KSQ was previously validated in English German and Dutch.

KSQ will be translated into Danish and validated in a Danish sarcoidosis population.

DETAILED DESCRIPTION:
KSQ will be linguistic validated according to existing guidelines. Consecutive patients with sarcoidosis will complete KSQ and other health questionnaires at baseline, after two weeks and 12 months. Concurrent validity, reliability, and responsiveness will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sarcoidosis
* Signed informed consent

Exclusion Criteria:

* Inability or unwillingness to adhere to the study
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish patients with sarcoidosis seen in Department of Respiratory Diseases Aarhus Denmark
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Internal consistency | At baseline
  Internal consistency, the interrelatedness of the items in the questionnaire, will be estimated by calculating Cronbach's α for each domain.
Test-retest reliability | At baseline
  Test-retest reliability will be evaluated by Intraclass correlation coefficients (ICC) and Bland- Altman plots comparing KSQ scores at baseline and at 14 days in stable patients
Concurrent validity | At baseline
  Concurrent validity was assessed by measuring the correlation of KSQ to other questionnaires
Responsiveness | 1 year from baseline
  Responsiveness:
  The ability to detect changes over time was assessed by measuring changes in KSQ over 12 months and correlating to changes in other questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Janne Møller, MD, Principal Investigator — AU
Locations (1):
- Aarhus University Hospital. Dep. of Respiatory Diseases and Allergology, Aarhus N, Denmark